CLINICAL TRIAL: NCT02043951
Title: A Prospective, Multicenter, Single Arm, Post-Market, Real-World Global Registry Assessing the Clinical Use and Safety of the LUTONIX Drug Coated Balloon Catheter in Arteries of the Lower Extremity (LUTONIX® Lower Extremity Global (LEG) Registry)
Brief Title: Use and Safety of the LUTONIX® Drug Coated Balloon Catheter in Arteries of the Lower Extremity
Acronym: LEG
Status: Terminated | Type: Observational
Why Stopped: Originally 500 patients were planned but only 59 have been enrolled
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: CL0015-01
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm: Lutonix Drug Coated Balloon
  Interventions: Device: Lutonix Drug Coated Balloon Catheter

INTERVENTIONS:
Device: Lutonix Drug Coated Balloon Catheter

SUMMARY:
The registry will enroll patients with claudication or critical limb ischemia and angiographically significant lesion(s) in arteries of the lower extremity. Subjects will be treated with the Lutonix® Drug Coated Balloon Catheter for approved indications according to the current country-specific Instructions for Use (IFU) and followed clinically for 1 year.

DETAILED DESCRIPTION:
This post-market registry is intended to assess the clinical use and safety of the Lutonix® Drug Coated Balloon Catheter in a heterogeneous patient population in real world clinical practice. Up to 500 patients will be enrolled in order to allow identification and assessment of rare adverse events (AEs) as well as outcomes in subpopulations defined by subject and lesion characteristics. All subjects will be followed for 1 year.

This registry is performed with marketed devices within the indications for use. There are no additional treatments or exams that will take place within this registry.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age;
2. Rutherford Clinical Category ≤ 5;
3. Patient or Legally Authorized Representative is willing to provide informed consent and comply with the required follow up;
4. Stenotic or obstructive vascular lesions in artery(s) of the lower extremity;
5. Lesion(s) can be treated with available LUTONIX Drug Coated Balloon Catheter device size matrix per current country-specific IFU.

Exclusion Criteria:

1. Patient is currently participating in an active phase of another investigational drug or device study;
2. Inability to take recommended medications as stated in the IFU or non-controllable allergy to contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world patients requiring drug coated balloon treatment.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Efficacy: Freedom from target lesion revascularization (TLR) | 12 months
Safety | 30 Days
  Freedom from the composite endpoint of target vessel revascularization (TVR), major amputation and major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of index limb and device- and procedure-related death.

SECONDARY OUTCOMES:
Acute Device Success | 30 days, 6 and 12 months
  Device success is defined as, a per device basis, the achievement of successful delivery and deployment of the registry device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the registry system. If a device is inserted into the subject but not used due to user error (e.g. inappropriate balloon length or transit time too long) this device will not be included in the device success assessment.
Procedural Success | 30 days, 6 and 12 months
  Attainment of ≤30% residual stenosis by visual estimate in the treatment area above the knee and attainment of ≤50% residual stenosis by visual estimate in the treatment area below the knee without major adverse events during the index procedure.
Freedom separately from each of the following adverse events listed below: | 30 days, 6 and 12 months
  * All-cause death
  * Device- and procedure-related mortality
  * Unexpected device or drug-related AEs
  * Index limb amputation (major and minor reported separately)
  * Reintervention for treatment of thrombosis of the target vessel
  * Reintervention for embolization to its distal vasculature
  * TLR (at 6 months)
  * TVR
  * Composite of all-cause perioperative (≤30 day) death and from the following: index limb amputation, index limb reintervention, and index-limb-related death
  * Major amputation and major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of index limb.

CONTACTS AND LOCATIONS:
Locations (8):
- The Vein Institute of Toronto, Toronto, Ontario, Canada
- Malaysia (4):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Universiti Kebangsaan, Kuala Lumpur
  - Hospital Universiti Sains Malaysia, Kubang Kerian Kelantan
  - Hospital Umum Sarawak, Sarawak
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Wellington Regional Vascular Centre, Newtown, Wellington
  - Tauranga Hospital, Tauranga